CLINICAL TRIAL: NCT02221323
Title: A Trial to Compare the Pharmacokinetics and Pharmacodynamics of Insulin Lispro Administered s.c. Into Lipohypertrophic or Normal Abdominal Adipose Tissue in Subjects With Diabetes Mellitus Type 1
Brief Title: A Trial to Compare the PK and PD of Insulin Lispro Administered Into Different Tissues in Subjects With Diabetes Mellitus Type 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DBC-14LIPOINJ01
Record Dates: First submitted 2014-08-15; First posted 2014-08-20 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin lispro (Experimental)
  Interventions: Drug: Insulin LISPRO

INTERVENTIONS:
Drug: Insulin LISPRO

SUMMARY:
The aim of this trial is to compare the pharmacokinetics and pharmacodynamics of insulin lispro injection into either lipohypertrophic lesions or normal tissue, utilizing both state-of-the-art euglycaemic clamp and mixed meal tolerance testing. The magnitude of insulin efficacy after injection into these different areas is still unclear. The results from this study may expand the knowledge on the severity of this issue and may provide evidence for future treatment recommendations regarding injection sites for insulin administration.

ELIGIBILITY:
Inclusion Criteria:

* AUCINS.0-4h and AUCGIR.0-4h during treatment period 1

Exclusion Criteria:

* AUCINS.0-4h and AUCBG.0-4h during treatment period 2, intra-subject variability of AUCINS.0-4h and AUCGIR.0-4h during treatment period 1

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
AUCINS.0-4h and AUCGIR.0-4h | up to 4 hours
  Compare the pharmacokinetic and pharmacodynamic effects of insulin lispro during the first 4 hours after s.c.
  administration into either lipohypertrophic or normal adipose tissue during a euglycaemic clamp examination.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Hövelmann, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, North Rhine-Westphalia, Germany